CLINICAL TRIAL: NCT00976287
Title: Autologous Bone Marrow Mesenchymal Stem Cells Transplantation Via Hepatic Artery in Patients With Liver Cirrhosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sun Yat-sen university, Sun Yat-sen university
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: zssy
Record Dates: First submitted 2009-08-31; First posted 2009-09-14 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Liver Cirrhosis
Keywords: Stem cells; Liver cirrhosis; Radiology; Interventional; Transplantation
MeSH Terms: conditions — Liver Cirrhosis | interventions — Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conserved Therapy (Active Comparator): Conserved Therapy
  Interventions: Procedure: Conserved Therapy
- Interventional Therapy (Experimental): Patients with liver cirrhosis were randomly separated into two groups. Autologous MSCs were infused to patients using interventional method via hepatic artery for One group. The catheter was inserted to proper hepatic artery. After the catheter placed at proper hepatic artery was confirmed by angiography, autologous bone marrow MSCs were infused slowly for 20-30 minutes. The control group accepted conserved therapy.
  Interventions: Procedure: Hepatic artery infusion

INTERVENTIONS:
Procedure: Hepatic artery infusion — Patients with liver cirrhosis were randomly separated into two groups. Autologous MSCs were infused to patients using interventional method via hepatic artery for One group. The catheter was inserted to proper hepatic artery. After the catheter placed at proper hepatic artery was confirmed by angiography, autologous bone marrow MSCs were infused slowly for 20-30 minutes. The control group accepted conserved therapy.
  Other Names: interventional therapy
  Arms: Interventional Therapy
Procedure: Conserved Therapy — Conserved Therapy
  Other Names: interventional; hepatic infusion
  Arms: Conserved Therapy

SUMMARY:
The purpose of this study is to investigate the efficacy of autologous bone marrow mesenchymal stem cells (MSCs) transplantation via hepatic artery in the treatment of liver cirrhosis. Liver function was monitored by serum examination. The levels of serum alanine aminotransferase (ALT), total bilirubin (TB), prothrombin time (PT) and albumin (ALB) were examined at pre-transplantation, and 3 days to 2 years post-transplantation. Child-Pugh scores and clinical symptoms were also observed simultaneously.

DETAILED DESCRIPTION:
Patients with liver cirrhosis were randomly separated into two groups. Autologous MSCs were infused to patients using interventional method via hepatic artery for One group. The catheter was inserted to proper hepatic artery. After the catheter placed at proper hepatic artery was confirmed by angiography, autologous bone marrow MSCs were infused slowly for 20-30 minutes. The control group accepted conserved therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years.
* Imaging evidences of liver cirrhosis.
* Child-Plough score of 10 or more.

Exclusion Criteria:

* Liver tumor on ultrasonography, CT or MRI examination.
* Problems in organs other than the liver(e.g.the heart or lungs).
* History of moderate to severe hepatic encephalopathy or variceal bleeding.
* Imaging evidences of vascular thromboses.
* Coma.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-01; Primary Completion 2009-12 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
The levels of serum alanine aminotransferase (ALT), total bilirubin (TB), prothrombin time (PT), albumin (ALB) | pre-transplantation, and 3 days to 2 years post-transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Zhu k shun, PHD, Study Director — SunYat-sen University